CLINICAL TRIAL: NCT01173640
Title: Resveratrol and Midazolam Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Bastyr University (Other)
Responsible Party: Principal Investigator, Yvonne Lin, Associate Professor, Pharmaceutics, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 38328
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: drug interactions; midazolam; cytochrome P450; resveratrol; pharmacokinetics
MeSH Terms: interventions — Midazolam; Resveratrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Midazolam Alone (Experimental): Baseline pharmacokinetics. On Study Visit Day 1, subjects will receive a single oral dose of midazolam (2 mg). Blood and urine will be collected to measure midazolam and its metabolites, and resveratrol and its metabolites.
  Interventions: Drug: Midazolam
- Single dose resveratrol (Experimental): On Study Visit Day 8, subjects will receive a 1 g oral dose of resveratrol followed 2 hours later by a single oral dose of midazolam (2 mg). Blood and urine will be collected to measure midazolam and its metabolites, and resveratrol and its metabolites.
  Interventions: Drug: Midazolam; Dietary Supplement: resveratrol (single dose)
- Multiple dose resveratrol (Experimental): Between Study Visit Days 8 and 15, subjects will take a 1 g dose of resveratrol daily. On Study Visit Day 15, subjects will receive a 1 g oral dose of resveratrol followed 2 hours later by a single oral dose of midazolam (2 mg). Blood and urine will be collected to measure midazolam and its metabolites, and resveratrol and its metabolites.
  Interventions: Drug: Midazolam; Dietary Supplement: resveratrol (multiple dose)

INTERVENTIONS:
Drug: Midazolam — 2 mg oral dose
  Other Names: Versed
Dietary Supplement: resveratrol (single dose) — 1 g oral dose
  Arms: Single dose resveratrol
Dietary Supplement: resveratrol (multiple dose) — 1 g oral dose for 8 days
  Arms: Multiple dose resveratrol

SUMMARY:
Adverse events due to drug-drug and/or herb-drug interactions are of serious concern and a major cause of morbidity and mortality. Resveratrol is a polyphenol antioxidant that has been identified in over 70 species and is suggested to be the constituent in red wine responsible for cardioprotective effects. The potential health benefits of resveratrol supplements are highly extolled in the alternative medicine industry and daily doses are up to 5 grams are being studied. While there are potential health benefits of high doses of resveratrol, for patients taking other drugs metabolized by CYP3A4, such as transplant medications, chemotherapies and HMG-CoA reductase inhibitors, there may be a clinically significant herb-drug interaction.

We, the investigators, have shown in vitro that resveratrol is a mechanism-based inhibitor of cytochrome P450 3A4 (CYP3A4). Based on our in vitro evidence and literature reports of the pharmacokinetics of resveratrol, we hypothesize that resveratrol will be a potent in vivo mechanism-based inhibitor of intestinal CYP3A4 enzymes. To date, there are no clinical studies that address the potential for a resveratrol-drug interaction. We propose to test whether single and multiple doses of resveratrol alter the pharmacokinetics of midazolam, a prototypic CYP3A4 probe drug.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years old.
* Body mass index between 18 and 30 kg/m2.
* Good health without a self-reported history of liver, kidney, gastrointestinal or heart disease
* Women use measures to avoid conception during the study period (e.g. oral contraceptives, intrauterine devices [IUDs], and condoms)
* Subjects must agree not to take any known substrates, inhibitors, inducers or activators of CYP3A4 at least 2 weeks before study start and for the entire duration of the study.
* Avoid ingesting grapefruit, grapefruit juice or other grapefruit juice containing products, and any herbal-based nutrient supplement or prescribed medications during the same period of time.
* Willing to fast overnight before the study days.
* Willing to abstain from alcohol-containing beverages 24 hours before and during the study visits, and willing to abstain from grapefruit, cranberry, blueberry products, peanuts and peanut butter, grape and grape products, and red wine at least one week prior to and during the study.

Exclusion Criteria:

* Current cigarette smoker
* Self-reported history of liver, kidney, gastrointestinal or heart disease
* Abnormal liver or kidney function tests based on the Comprehensive and Hepatic Panel (below the lower end or greater than 15% of the upper end of the reference range).
* Known or suspected history of alcohol or drug abuse
* Allergic to benzodiazepines or any other chemically related drugs
* Women who are pregnant or breastfeeding
* Recent ingestion (<1 week) of any medication known to be metabolized by CYP3A4 or alter CYP3A activity
* Chronic use of prescription drugs, over-the-counter, vitamins or natural products. However, oral contraceptives will be permitted.
* Unable to give informed consent
* Participated in another clinical trial or study within 30 days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Inhibition of midazolam clearance | 3 study visit days
  The primary aim will be to determine if resveratrol causes inhibition of intestinal and hepatic CYP3A4 enzymes as determined by oral midazolam clearance following single and multiple doses of resveratrol, respectively.

SECONDARY OUTCOMES:
Resveratrol accumulation | 3 study visit days
  Secondary aims will be to measure circulating levels of resveratrol and its conjugated metabolites following single and multiple doses of resveratrol and to determine resveratrol accumulation in low density lipoproteins (LDL).

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne S Lin, PhD, Principal Investigator — University of Washington; Ryan Bradley, ND, MPH, Principal Investigator — Bastyr University; Kelsey Hanson, MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States